CLINICAL TRIAL: NCT00979238
Title: An Open Label Dose-Escalation Study Of A Self Complementary Adeno-Associated Viral Vector (scAAV 2/8-LP1-hFIXco) For Gene Transfer in Hemophilia B
Brief Title: Dose-Escalation Study Of A Self Complementary Adeno-Associated Viral Vector For Gene Transfer in Hemophilia B
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Hemophilia of Georgia, Inc. (Other); Children's Hospital of Philadelphia (Other); University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AGT4HB; 5R01HL094396 (NIH)
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Hemophilia B
Keywords: Hemophilia B; Factor IX Gene; Factor IX Protein; Vector
MeSH Terms: conditions — Hemophilia B | interventions — Genetic Engineering; Disease Vectors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Group 1 (Other): All participants who meet the eligibility requirements.
  Intervention: Gene Transfer and drug (scAAV2/8-LP1-hFIXco).
  Interventions: Genetic: Gene Transfer; Drug: scAAV2/8-LP1-hFIXco

INTERVENTIONS:
Genetic: Gene Transfer — Peripheral vein infusion of scAAV2/8-LP1-hFIXco vector once per participant
Drug: scAAV2/8-LP1-hFIXco — Peripheral vein infusion of scAAV2/8-LP1-hFIXco vector once per participant.
  Other Names: vector

SUMMARY:
The purpose of this study is to determine the safety of giving a normal factor IX gene to treat individuals who have an abnormal or no factor IX gene. Recruitment will be limited to adults (≥ 18 years) with a confirmed diagnosis of hemophilia B (HB), resulting from a missense mutation in the coagulation factor IX (FIX) gene or a nonsense mutation that has not been associated with an inhibitor. Only subjects who have no evidence of active hepatitis or anti-hFIX antibodies, and who have been treated/exposed to Factor IX concentrates for at least ten years and have had an average of 3 bleeding episodes per year requiring FIX administration will be enrolled. Patients will be recruited within the United States for treatment at St. Jude Children's Research Hospital, and patients will be recruited in England and other countries for treatment in London by our British collaborators.

DETAILED DESCRIPTION:
Hemophilia B is caused by an absence or abnormality in the gene that produces the factor IX protein. Affected individuals cannot make a blood clot effectively and suffer from severe bleeding episodes. Repeated bleeding episodes, specifically into joints, can cause chronic joint disease and lead to disability. This research study will test the safety of giving an affected individual a normal factor IX gene which can produce factor IX protein in his body. We will give the normal gene for factor IX by using an inactivated (not able to function) virus called "the vector." The vector used in this study was developed from an adeno-associated virus that has been changed so that it is unable to cause a viral infection in humans. This inactivated virus was further altered to carry the factor IX gene and to locate within liver cells where factor IX protein is normally made.

The protocol long-term follow-up (LTFU) period was changed from 15 years to 5 years in accordance with the FDA guidance for participants who received human gene therapy products. The FDA updated the guidance stating their current recommendations for the duration of an LTFU protocol, based on product, to be up to five years for AAV vectors.

All study participants have completed 5 years of follow-up and are being transitioned off study.

ELIGIBILITY:
Inclusion Criteria:

* Males ≥ 18 years of age with established severe HB (FIX:C<1u/dl),
* Treated/exposed to FIX products (e.g., concentrates or fresh frozen plasma) for at least 10 years or 50 exposure days.
* A minimum of an average of 3 bleeding episodes per year requiring FIX infusions or prophylactic FIX infusions because of frequent prior bleeding episodes
* Able to give informed consent and comply with requirements of the trial
* Currently free of inhibitor and have no history of inhibitors to FIX protein
* A negative family history for the development of an inhibitor,
* Willing to practice a reliable barrier method of contraception until 3 sequential samples are negative for vector genomes using our PCR assay.

Exclusion Criteria:

* Evidence of active infection with Hepatitis B or C virus as reflected by HBsAg or NCV RNA positivity, respectively. To be considered negative for active infection, two negative assays at a minimum of a six month interval are required.
* Exposure to Hepatitis B or C who are currently on antiviral therapy.
* Serological evidence of HTLV or active HIV infection. Individuals who are effectively being treated with antiretroviral therapy are eligible. Specific criteria for effectiveness of treatment include the following:

  * Documented CD4+ T-cell count of > 350 cells/mm^3.
  * HIV-1 RNA viral load < 400 copy/ml for at least the past 12 months, including at least 2 viral load test results of < 400 copy/ml during the immediate 12 month interval prior to screening.
  * Screening HIV-RNA viral load < 400 copies/ml.
  * Stable HAART regimen (drugs of at least 2 different classes) for at least 12 months prior to study entry. Treatment regimen changes for dosing convenience and in response to toxicity are permitted.
  * Documented and confirmed (repeated) viral loads of ≥ 400 copies/ml during the 12 month time interval prior to screening are bases for exclusion although a single, unconfirmed, "glimpse" of ≥ 400 copies/ml are permitted.
* Significant liver dysfunction as defined by an abnormal ALT (alanine transaminase), bilirubin, alkaline phosphatase or INR. Potential participants who have had a liver biopsy in the past 3 years will be excluded if they have significant fibrosis of 3 or 4 as rated on a scale of 0-4.
* Coronary artery disease as a co-morbid condition
* Platelet count of <50 x 10^9/l
* Creatinine ≥ 1.5 mg/dl
* Hypertension with systolic blood pressure (BP) ≥ 140 mmHg or diastolic BP ≥ 90 mmHg
* History of active tuberculosis, fungal disease or other chronic infection
* History of chronic disease that would adversely affect performance other than hemophilic arthropathy
* Detectable antibodies reactive with AAV8
* Subjects who are unwilling to provide the required semen samples
* Poor performance status (WHO performance status score >1) or
* Received an AAV vector or any other gene transfer agent in the previous 6 months
* Presence of lung nodule(s) suspicious of malignancy on screening chest tomography
* Presence of liver abnormalities suspicious of malignancy on screening liver ultrasound

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-02-22 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of systemic administration of a novel self-complementary AAV vector in adults with severe hemophilia B at up to four different dosage levels. | 15 years
  Outcome measures are descriptive in nature but data collected in a longitudinal manner will also be analyzed (as and when appropriate) using longitudinal methods such as mixed effect model which takes into account the correlation among the observation taken at various time points within a participant.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Reiss, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (8):
- United States (7):
  - Stanford Medical School, Stanford, California
  - University of Kentucky, Lexington, Kentucky
  - Oregon Health and Science University, Portland, Oregon
  - Hemophilia Center of Western Pennsylvania, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - Scott and White Memorial Hospital, Temple, Texas
- Katharine Dormandy Haemophilia Centre and Haemostasis Unit, University College of London, London, United Kingdom

REFERENCES:
- [Derived] Reiss UM, Davidoff AM, Tuddenham EGD, Chowdary P, McIntosh J, Muczynski V, Journou M, Simini G, Ireland L, Mohamed S, Riddell A, Pie AJ, Hall A, Quaglia A, Mangles S, Mahlangu J, Haley K, Recht M, Shen YM, Halka KG, Fortner G, Morton CL, Gu Z, Hayden RT, Neufeld EJ, Okhomina VI, Kang G, Nathwani AC. Sustained Clinical Benefit of AAV Gene Therapy in Severe Hemophilia B. N Engl J Med. 2025 Jun 12;392(22):2226-2234. doi: 10.1056/NEJMoa2414783. PMID 40499172
- [Derived] Nathwani AC, Reiss UM, Tuddenham EG, Rosales C, Chowdary P, McIntosh J, Della Peruta M, Lheriteau E, Patel N, Raj D, Riddell A, Pie J, Rangarajan S, Bevan D, Recht M, Shen YM, Halka KG, Basner-Tschakarjan E, Mingozzi F, High KA, Allay J, Kay MA, Ng CY, Zhou J, Cancio M, Morton CL, Gray JT, Srivastava D, Nienhuis AW, Davidoff AM. Long-term safety and efficacy of factor IX gene therapy in hemophilia B. N Engl J Med. 2014 Nov 20;371(21):1994-2004. doi: 10.1056/NEJMoa1407309. PMID 25409372
- [Derived] Nathwani AC, Tuddenham EG, Rangarajan S, Rosales C, McIntosh J, Linch DC, Chowdary P, Riddell A, Pie AJ, Harrington C, O'Beirne J, Smith K, Pasi J, Glader B, Rustagi P, Ng CY, Kay MA, Zhou J, Spence Y, Morton CL, Allay J, Coleman J, Sleep S, Cunningham JM, Srivastava D, Basner-Tschakarjan E, Mingozzi F, High KA, Gray JT, Reiss UM, Nienhuis AW, Davidoff AM. Adenovirus-associated virus vector-mediated gene transfer in hemophilia B. N Engl J Med. 2011 Dec 22;365(25):2357-65. doi: 10.1056/NEJMoa1108046. Epub 2011 Dec 10. PMID 22149959
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols